CLINICAL TRIAL: NCT04780646
Title: Effects of Urban Nature on Stress and Quality of Life of Subjects With Elevated Stress Levels - a Three-armed Randomized Controlled Study
Brief Title: Effects of Urban Nature on Stress and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stadtnatur
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Stress, Psychological
Keywords: Nature therapy; Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nature therapy in urban nature (Experimental): Subjects receive a 90-minute nature therapy session once per week for 8 weeks with a licensed nature therapist, who explains exercises on perceiving nature and the connection between nature and health.
  Interventions: Behavioral: Nature therapy in urban nature
- City Walk (Active Comparator): Subjects receive a 90-minute city walk through urban sourroundings once per week for 8 weeks with a city guide, who talks about city architecture and gives information about the history of the surroundings.
  Interventions: Behavioral: City Walk
- Waiting List (No Intervention): Subjects don't receive any therapy.

INTERVENTIONS:
Behavioral: Nature therapy in urban nature — Nature therapy means visits in nature, actively perceiving the flora and fauna
  Arms: Nature therapy in urban nature
Behavioral: City Walk — City Walk means walking through urban surroundings (houses, streets, concrete..) with as little as possible contact to nature
  Arms: City Walk

SUMMARY:
The aim of this study is to investigate the effects of regular nature therapy in urban nature with guidance of a licensed nature therapist on stress, quality of life and physical symptoms of subjects with elevated stress levels.

ELIGIBILITY:
Inclusion Criteria:

* stress with at least 4 of 10 points on the Numeric Analogue Scale (NAS) at least 1 month
* at least 3 of the following 8 stress-associated symptoms: sleep disturbances, inappetence or increased appetite, shoulder neck tension/back pain, tension headache, concentration disturbances, exhaustion, nervousness/irritability, stress-associated digestive complaints.

Exclusion Criteria:

* serious acute or chronic diseases
* pregnancy or lactation
* known serious mental illness
* immobility or restriction for gymnastics exercises due to orthopaedic, neurological or other medical cause
* participation in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items while higher values meaning a higher grade of perceived stress.

SECONDARY OUTCOMES:
Zerssen symptom list (B-LR and B-LR') | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 20-80, higher score meaning a better outcome
International Physical Activity Questionnaire (IPAQ) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  MET minutes represent the amount of energy expended carrying out physical activity. To get a continuous variable score from the IPAQ (MET minutes a week) we will consider walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS; higher score meaning better outcome; range 0 to around 3000 MET minutes a week
Maslach Burnout Inventory (MBI) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 0-96, higher score meaning a better outcome
Mindfulness (Freiburger Fragebogen zur Achtsamkeit, FFA) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 0-56, higher score meaning a better outcome
General Self-Efficacy Short Scale-3 (GSE-3) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
Perceived Benefits of Nature Questionnaire (PBNQ) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  mean score of the 11 items, range 1-7, lower score meaning a better outcome
Subjective Vitality Scale (SVS-G state) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range from 0-28, lower score meaning a better outcome
Flourishing Scale (FS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Assessing full scale, range 8-56, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
Profile of Mood States (POMS) | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
Sociodemographic Measurements | Date of Inclusion (Baseline)
  Age, gender, marital status, number of people in household, education level, employment status, job, personal net income, household income
Behavioural questions: doctor visits and health | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  amount of doctor visits, amount of sick leave days in the last 2 months
Expectation questions | Date of Inclusion (Baseline)
  for intervention 1 and 2 on a 6-point likert scale from 1 (very strong) to 6 (nothing at all)
Behavioural questions: cigarette consumption | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Number of cigarettes on average per day in the last month
Behavioural questions: alcohol consumption | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  Number of alcoholic beverages on average per week in the last month
Behavioural questions: time in nature | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  amount of hours spent in nature per week in the last month
Behavioural questions: nature as priority | Date of Inclusion (Baseline), after 8 weeks and after 16 weeks
  if spending time in nature is seen as a priority on a 6-point likert scale 1 (very strong) to 6 (nothing at all)
Heart Rate (HR) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by faros 180
Heart Rate Variability (HRV) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by faros 180

OTHER OUTCOMES:
Qualitative interviews in individual interviews | 8 weeks after inclusion
  Qualitative assessment will be carried out in 45-minute individual interviews in 20 (randomized selected) patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus
Locations (1):
- Charite University, Berlin, Germany